CLINICAL TRIAL: NCT03284112
Title: Old SCHOOL Hip-Hop: A Randomized Controlled Trial to Improve Alzheimer's Disease Knowledge
Brief Title: Old SCHOOL Hip-Hop: Improve Alzheimer's Disease Knowledge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, James M Noble, MD, MS, CPH, FAAN, Professor of Neurology in the Taub Institute and the Sergievsky Center, Department of Neurology - Aging & Dementia, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAR5473; 5R01AG054536 (NIH)
Record Dates: First submitted 2017-09-12; First posted 2017-09-15 (Actual); Results first posted 2025-10-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Dementia
Keywords: Dementia, Schools, Nutrition, Health
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): School population without the Old SCHOOL Hip-Hop program, but with the My Plate program.
  Interventions: Behavioral: My Plate
- Intervention (Experimental): School population with the Old SCHOOL Hip-Hop program.
  Interventions: Behavioral: Old SCHOOL Hip-Hop

INTERVENTIONS:
Behavioral: Old SCHOOL Hip-Hop — A school-based intervention called "Old S.C.H.O.O.L. Hip-Hop" (OSHH) or Seniors Can Have Optimal aging and Ongoing Longevity, to educate 4th and 5th grade students (ages 9-11y) about key dementia signs and symptoms, basic pathophysiology of Alzheimer disease, and the importance of early recognition, care-seeking behavior, and preventative measures (lifelong healthy lifestyle decisions). The intervention is delivered in a classroom or school auditorium setting, using an innovative, modular, multimedia program and home-based activities, to increase parental and family dementia literacy.
  Other Names: OSHH Program
  Arms: Intervention
Behavioral: My Plate — The program selected for the control arm, "My Plate," will address nutrition, physical activity, and obesity education. This program was selected because nutrition, physical activity, and wellness programs are now being incorporated into New York City public school curriculums as part of a legislative directive. Trained facilitators will conduct "My Plate" as an entry point for the USDA's My Plate nutrition program. Students will learn about My Plate across the 3-day one-hour-a-day program.
  Other Names: My Plate nutrition program
  Arms: Control

SUMMARY:
The purpose of this research study is to evaluate the knowledge of parents and children with respect to dementia symptoms, risk factors, and response before and after an interactive dementia education program that uses music and dance to enhance a health education curriculum at 1-week and 3-months after the intervention.

DETAILED DESCRIPTION:
Public awareness of cardinal Alzheimer's disease (AD) symptoms remains low. Adults often underestimate personal dementia risk; minority populations are more likely to have low dementia literacy and be unaware of it. Cultural dementia belief in minority groups are complex and pose barriers to diagnosis, with dementia symptoms being considered a part of normal aging, or that discussion may be taboo even when recognized. A key barrier to timely AD diagnosis in African Americans is delayed physician contact, often years-long, following the onset of first symptoms. Despite studies demonstrating that dementia concepts first develop in elementary school periods, apart from our work, no dementia awareness programs focus on children. This intervention therefore addresses a major gap regarding optimal approaches for shifting cultural perceptions of dementia in low-income minority populations and reducing barriers to its timely diagnosis.

All R01 aims have been completed in this study.

ELIGIBILITY:
Inclusion Criteria:

* 4th and 5th-grade children (ages 9-11y) and their parents (age > 20 years).
* Selected New York City public schools with similar socio-demographic composition.

Exclusion Criteria:

* Schools have already received pilot OSHH and the U.S. Department of Health and Human Services (HHS) programming.

Min Age: 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2244 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Noble, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: NYC schools were recruited & enrolled from September 9, 2018 through February 27, 2023. Once each school agreed to participate, parents & students were recruited. Then each school was randomized into either Control or Intervention arm.
Units Other Than Participants: Schools
Groups:
- Control Students & Parents: School & parent population without the Old SCHOOL Hip-Hop program, but with the My Plate program.
  My Plate: The program selected for the control arm, "My Plate," will address nutrition, physical activity, and obesity education. This program was selected because nutrition, physical activity, and wellness programs are now being incorporated into New York City public school curriculums as part of a legislative directive. Trained facilitators will conduct "My Plate" as an entry point for the USDA's My Plate nutrition program. Students will learn about My Plate across the 3-day one-hour-a-day program.
- Intervention Students & Parents: School & parent population with the Old SCHOOL Hip-Hop program.
  Old SCHOOL Hip-Hop: A school-based intervention called "Old S.C.H.O.O.L. Hip-Hop" (OSHH) or Seniors Can Have Optimal aging and Ongoing Longevity, to educate 4th and 5th grade students (ages 9-11y) about key dementia signs and symptoms, basic pathophysiology of Alzheimer disease, and the importance of early recognition, care-seeking behavior, and preventative measures (lifelong healthy lifestyle decisions). The intervention is delivered in a classroom or school auditorium setting, using an innovative, modular, multimedia program and home-based activities, to increase parental and family dementia literacy.
Period: Overall Study
Arm/Group | Control Students & Parents | Intervention Students & Parents
Started | 1175; 14 Schools | 1069; 14 Schools
Parents Started | 401; 14 Schools | 382; 14 Schools
Children Started | 774; 14 Schools | 687; 14 Schools
Parents Completed | 344; 14 Schools | 349; 14 Schools
Children Completed | 741; 14 Schools | 665; 14 Schools
Completed | 1085; 14 Schools | 1014; 14 Schools
Not Completed | 90; 0 Schools | 55; 0 Schools

BASELINE CHARACTERISTICS:
Groups:
- Control Students: School population without the Old SCHOOL Hip-Hop program, but with the My Plate program.
  My Plate: The program selected for the control arm, "My Plate," will address nutrition, physical activity, and obesity education. This program was selected because nutrition, physical activity, and wellness programs are now being incorporated into New York City public school curriculums as part of a legislative directive. Trained facilitators will conduct "My Plate" as an entry point for the USDA's My Plate nutrition program. Students will learn about My Plate across the 3-day one-hour-a-day program.
- Intervention Students: School population with the Old SCHOOL Hip-Hop program.
  Old SCHOOL Hip-Hop: A school-based intervention called "Old S.C.H.O.O.L. Hip-Hop" (OSHH) or Seniors Can Have Optimal aging and Ongoing Longevity, to educate 4th and 5th grade students (ages 9-11y) about key dementia signs and symptoms, basic pathophysiology of Alzheimer disease, and the importance of early recognition, care-seeking behavior, and preventative measures (lifelong healthy lifestyle decisions). The intervention is delivered in a classroom or school auditorium setting, using an innovative, modular, multimedia program and home-based activities, to increase parental and family dementia literacy.
- Control Parents: Parents of school population without the Old SCHOOL Hip-Hop program, but with the My Plate program.
  My Plate: The program selected for the control arm, "My Plate," will address nutrition, physical activity, and obesity education. This program was selected because nutrition, physical activity, and wellness programs are now being incorporated into New York City public school curriculums as part of a legislative directive. Trained facilitators will conduct "My Plate" as an entry point for the USDA's My Plate nutrition program. Students will learn about My Plate across the 3-day one-hour-a-day program.
- Intervention Parents: Parents of school population with the Old SCHOOL Hip-Hop program. Old SCHOOL Hip-Hop: A school-based intervention called "Old S.C.H.O.O.L. Hip-Hop" (OSHH) or Seniors Can Have Optimal aging and Ongoing Longevity, to educate 4th and 5th grade students (ages 9-11y) about key dementia signs and symptoms, basic pathophysiology of Alzheimer disease, and the importance of early recognition, care-seeking behavior, and preventative measures (lifelong healthy lifestyle decisions). The intervention is delivered in a classroom or school auditorium setting, using an innovative, modular, multimedia program and home-based activities, to increase parental and familv dementia literacy.
- Total: Total of all reporting groups
Arm/Group | Control Students | Intervention Students | Control Parents | Intervention Parents | Total
Number analyzed (Participants) | 774 | 687 | 401 | 382 | 2244
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 774 | 687 | 0 | 0 | 1461
  18-64 years | 0 | 0 | 387 | 369 | 756
  >=65 years | 0 | 0 | 4 | 6 | 10
  Unknown/Not Reported | 0 | 0 | 10 | 7 | 17
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 362 | 374 | 354 | 325 | 1415
  Male | 334 | 274 | 42 | 47 | 697
  Unknown/Not Reported | 78 | 39 | 5 | 10 | 132
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 17 | 9 | 19 | 9 | 54
  Native Hawaiian or Other Pacific Islander | 3 | 0 | 3 | 0 | 6
  Black or African American | 158 | 214 | 209 | 232 | 813
  White | 52 | 38 | 54 | 43 | 187
  Unknown/Not Reported (Other) | 544 | 426 | 116 | 98 | 1184
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 106 | 87 | 118 | 97 | 408
  Not Hispanic | 218 | 245 | 268 | 267 | 998
  Unknown | 450 | 355 | 15 | 18 | 838
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 774 | 687 | 401 | 382 | 2244
Baseline Alzheimer's Disease Knowledge Using ASK-AD 7 [Mean (Standard Deviation); unit: units on a scale] — Baseline Knowledge of Alzheimer's Disease using 7-item scale: ASK-AD 7 (Assess Symptoms and Knowledge of Alzheimer's Disease - 7 Questions). Minimum value is 0 and maximum value is 7. Higher scores indicate greater number of questions answered correctly, indicating a better outcome. Population: Each row indicates parents & students which were treated as two separate groups. The number of parents + number of students who completed a baseline measure = overall population.
  units on a scale
    Students Pre-Test: Immediately Before Intervention: number analyzed (Participants) | 774 | 687 | 0 | 0 | 1461
    Students Pre-Test: Immediately Before Intervention | 2.98 (1.93) | 2.75 (1.97) |  |  | 2.87 (1.95)
    Parents Pre-Test: Before Intervention: number analyzed (Participants) | 0 | 0 | 401 | 382 | 783
    Parents Pre-Test: Before Intervention |  |  | 5.13 (1.77) | 5.24 (1.70) | 5.18 (1.74)

OUTCOME MEASURES:

1. Primary Outcome: OSHH Program Effectiveness of Educating Parents at 1-week and 3-months After the Intervention Using ASK-AD 7
Description: OSHH Program effectiveness of educating parents at 1-week post and 3-months post intervention using a 7-item scale: ASK-AD 7 (Assess Symptoms and Knowledge of Alzheimer's Disease - 7 Questions). Minimum value is 0 and maximum value is 7. Higher scores indicate greater number of questions answered correctly, indicating a better outcome.
Time Frame: Baseline (1 week up to 15 weeks prior to Intervention Day 1), 1-week post-intervention (1 week up to 13 weeks post-Intervention Day 3, but always before 3-month intervention), and 3-months post-intervention (10 to 24 weeks post-intervention Day 1)
Population: Parents whose children participated in either Control Arm (MyPlate Program) or Intervention Arm (Old School Hip Hop Program) and who consented to participate in the survey.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 401 | 382
score on a scale
  Pre-Test (1 week prior to intervention) | 5.14 (0.09) | 5.28 (0.08)
  Post-Test (1-week post intervention) | 5.41 (0.08) | 5.62 (0.07)
  Delayed Post-Test (3-months post intervention) | 5.68 (0.09) | 5.95 (0.09)

2. Secondary Outcome: OSHH Program Effectiveness of Educating Students at Immediate-post and 3-months Post the Intervention Using ASK-AD 7
Description: OSHH Program effectiveness of educating students immediately-post and 3-months post the intervention using a 7-item scale: ASK-AD 7 (Assess Symptoms and Knowledge of Alzheimer's Disease - 7 Questions). Minimum value is 0 and maximum value is 7. Higher scores indicate greater number of questions answered correctly, indicating a better outcome.
Time Frame: Immediately before intervention began (On Day 1 of programming), Immediately post intervention (Day 3 of programming), 3-months post intervention (6 up to 20 weeks post Day 1 of programming)
Population: Students randomized into either Control Arm (My Plate program) or Intervention Arm (Old School Hip Hop program)
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Control: Students: School population without the Old SCHOOL Hip-Hop program, but with the My Plate program.
  My Plate: The program selected for the control arm, "My Plate," will address nutrition, physical activity, and obesity education. This program was selected because nutrition, physical activity, and wellness programs are now being incorporated into New York City public school curriculums as part of a legislative directive. Trained facilitators will conduct "My Plate" as an entry point for the USDA's My Plate nutrition program. Students will learn about My Plate across the 3-day one-hour-a-day program.
- Intervention: Students: School population with the Old SCHOOL Hip-Hop program.
  Old SCHOOL Hip-Hop: A school-based intervention called "Old S.C.H.O.O.L. Hip-Hop" (OSHH) or Seniors Can Have Optimal aging and Ongoing Longevity, to educate 4th and 5th grade students (ages 9-11y) about key dementia signs and symptoms, basic pathophysiology of Alzheimer disease, and the importance of early recognition, care-seeking behavior, and preventative measures (lifelong healthy lifestyle decisions). The intervention is delivered in a classroom or school auditorium setting, using an innovative, modular, multimedia program and home-based activities, to increase parental and family dementia literacy.
Arm/Group | Control: Students | Intervention: Students
Number analyzed (Participants) | 774 | 687
score on a scale
  Pre-test (Immediately Before Intervention) | 3.13 (0.18) | 3.36 (0.18)
  Post-Test (Immediately Post Intervention) | 3.67 (0.17) | 5.02 (0.17)
  Delayed Post-Test (3-months post intervention) | 4.21 (0.18) | 6.69 (0.18)

ADVERSE EVENTS:
Time Frame: Through study completion, up to 24 weeks.
Description: Undue psychological burden on child or child being upset due to discussing Alzheimer's Disease
Arm/Group | Control Students | Intervention Students | Control Parents | Intervention Parents
All-Cause Mortality (participants affected / at risk) | 0/774 | 0/687 | 0/401 | 0/382
Serious Adverse Events (participants affected / at risk) | 0/774 | 0/687 | 0/401 | 0/382
Other Adverse Events (participants affected / at risk) | 0/774 | 0/687 | 0/401 | 0/382

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-16): https://cdn.clinicaltrials.gov/large-docs/12/NCT03284112/Prot_SAP_000.pdf